CLINICAL TRIAL: NCT05026242
Title: Effects of Almond Consumption on Innate Myeloid and Lymphoid Cells Composition and Activity
Brief Title: Effects of Almond Consumption on Innate and Adaptive Immune System
Acronym: AlmondIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IH-21-BULLOM-NR-01
Record Dates: First submitted 2021-07-15; First posted 2021-08-30 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Immune System
Keywords: almonds; innate myeloid; lymphoid cells; immune function; miRNAs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond intervention (Experimental): Participants will follow their regular Western-style diet substituting unhealthy snacks by 2-daily servings of almonds
  Interventions: Behavioral: Almond intervention
- Control (Active Comparator): Participants will be provided with isocaloric snacks
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Almond intervention — Participants will follow their regular Western-style diet substituting unhealthy snacks by 2-daily servings of almonds
  Arms: Almond intervention
Behavioral: Control — Participants will be provided with isocaloric snacks
  Arms: Control

SUMMARY:
Almonds are a rich matrix of different nutrients with demonstrated benefits on immune system. This proposal examines the effect of regular consumption of almonds on innate and adaptive immune system in healthy individuals with overweight regularly consuming a Western-style diet and unhealthy snacks.

DETAILED DESCRIPTION:
In the last months, with the whole world grappling with COVID-19 and because like in many other diseases, the host immune system determines the progress of COVID-19 and the severity, there is a frantic race for finding treatment strategies based on current knowledge until effective vaccine is developed. Therefore, the modulation of inflammatory response and cytokine production using immunonutrition makes more sense than ever.

The almond is a tree nut, rich in fiber, vitamin E, biotin, minerals such as magnesium and phytonutrients, specifically flavonoids, plant sterols, phenolic acids and could have a potential beneficial role in immune system. However, beyond its beneficial role and down-lowering specific circulating cytokines in low-grade chronic inflammatory diseases, the role of almond on both innate and adaptive immune system has not been explored.

The investigators hypothesize that regular consumption of almonds will contribute to strengthening the immune system through the modulation of specific circulating miRNAs.

The primary objective is to evaluate the effect of almond consumption on the maturation of innate lymphoid cells (ILCs).

Secondarily, the insvestigators aims to:

1. Examine the effect of regular consumption of almonds in the context of a Western-style diet on: a) innate immune system through the analysis of other blood cell populations including monocytes and lymphocyte's subsets (T-cells, B-cells). b) adaptive immune system assessed by: b.1) circulating inflammatory markers and b.2) ex-vivo ability for peripheral blood mononuclear cell (PBMC) to produce cytokines.

   c) circulating miRNAs, focusing in immune-related miRNAs.
2. To investigate whether changes in miRNAs mediate the effect of almonds on ILCs activity and the other innate and adaptive immune system indicators analysed.

The expected results would enhance understanding of the role of almonds in immune function, to establish the basis of new research for the promotion of the health benefits of nuts in immune-related diseases and facilitate the use of personalized nutrition to improve human health.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25.0-34.9 Kg/m2
* Western-style diet
* Unhealthy snacks other than nuts (i.e. potato chips, crackers, corn puffs, pretzels, pastries, cookies, candies) >1 serving/day

Exclusion Criteria:

* Regular smokers (≥ 10 cigarettes/day)
* Diagnoses of type 2 diabetes
* Cardiovascular disease, chronic kidney disease, liver disease, active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption, cancer - active malignant cancer or history of malignancy within the last 5 years, psychiatric disorders
* Use of anti-inflammatory or antioxidants drugs
* Not stable medication in the last 3 months
* Regular alcohol consumption above of the national recommendations or drug abuse
* Frequent consumption of nuts
* Allergy to the intervention products or other severe allergies and food intolerances
* Dietary patterns interfering with the study protocol (e.g. vegetarian, vegan, low carbohydrate dieters, high fat dieters) two months prior inclusion, during the study or plans to initiate during the study
* Daily use of multivitamin or mineral supplements
* Bad dentures, implying difficulty to chew nut
* Pregnancy or lactation, pregnancy within the past 12 month or plans to become pregnant during the study
* Consumption of probiotics or prebiotics in the last 3 months and laxatives

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in innate myeloid and lymphoid cells | These outcomes will be assessed at baseline and at 8 weeks
  CD45+, CD103+, CD56+, CD14+,CD16+, CD8+, CD19+, CD4+, CD3+, CD36+, CD44+, ROR γ t, NKp46+, FoxP3+ will be assessed by means of flow cytometry in cryopreserved cells.

SECONDARY OUTCOMES:
Changes in lymphocyte subsets | These outcomes will be assessed at baseline and at 8 weeks
  Lymphocyte subsets will be measured using Ficoll-Paque (GE Healthcare) density gradient centrifugation and flow cytometry. Results will be expressed in 10 (9)/L cells
Changes in immune cells activity assessed by citokyne production | These outcomes will be assessed at baseline and at 8 weeks
  Innate lymphoid and myeloid cells activity will be assessed in cryopreserved PBMCs. Inflammation mediators ( such as hs-CRP, IL1, IL2, IL4, IL-6, IL-7, IL-10, TNFα, IFN-γ, TGF-β, TLR4, NOD1) will be assessed with chemical assays (ELISA). Results will be expressed as mass/volume
Changes in immune cells activity assessed by adaptor molecules | These outcomes will be assessed at baseline and at 8 weeks
  A study of the molecular signaling using Western blot qauntification of adaptor molecules that play a pivotal role in immune cell activation through Toll-like receptors and therefore are good markers for specific immune cells activities
Changes in inflammatory markers and related molecules in plasma/serum | These outcomes will be assessed at baseline and at 8 weeks
  Several citokynes related immune cells (i.e TNF, IL6, IL1) and other circulating inflmmatory markers (i.e. CRP, amiloid) will be measured by ELISA related methods. Results will be expressed in mass/volume

OTHER OUTCOMES:
Changes in circulating miRNAs | These outcomes will be assessed at baseline and at 8 weeks
  20 circulating miRNA will be measured using TaqMan MicroRNA Assays. Results will be expressed as relative increase or decrease
Changes in gut microbiota composition | These outcomes will be assessed at baseline and at 8 weeks
  16S RNA will be sequenced and functional in silico analyses using existing datasets will be conducted. Data will be expressed in relative abundace (OTUS/ASV) at genus, family and/or specie level
Changes in gut microbiota function | These outcomes will be assessed at baseline and at 8 weeks
  Fecal targeted quantitative metabolomic multi-platform analyses will be conducted to identify changes in fecal metabolites related to the intervention (different metabolites including lipid species, aminoacids, bile acids, short-chain fatty acids...will be included)
Changes in circulating metabolites concentrations | These outcomes will be assessed at baseline and at 8 weeks
  We will use a multi-platform targeted/untargeted approach to identify/quantify metabolites related to the intervention and outcomes. (different metabolites including lipid species, aminoacids, bile acids, short-chain fatty acids...will be included)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bullo, Prof, Principal Investigator — Pere Virgili
Locations (1):
- IISPV, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No
Data sharing will be upon request directly to the PI